CLINICAL TRIAL: NCT00437008
Title: Acute Effects of a Low-AGE vs. High-AGE Meal on Postprandial Endothelial Function in People With Type 2 Diabetes Mellitus. Protective Effects of Benfotiamine
Brief Title: Effects of Benfotiamine and AGE on Endothelial Function in People With Diabetes
Acronym: AGE-Benfo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Benfo-1-2005
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Endothelial Dysfunction; Type 2 Diabetes Mellitus
Keywords: endothelial dysfunction; flow-mediated dilatation; advanced glycation end products; postprandial
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — benphothiamine

INTERVENTIONS:
Drug: Benfotiamine 1050mg, 3 days
Behavioral: high-AGE vs. low-AGE meal

SUMMARY:
The purpose of the study is to determine whether there are differences in postprandial endothelial function following a high-AGE(Advanced Glycation End-products) meal vs. a low-AGE meal. We also intend to investigate if the therapy with 1050mg Benfotiamine for 3 days protects against the postulated deterioration of endothelial function after a high-AGE meal in people with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
AGEs are a heterogeneous group of compounds formed by the nonenzymatic reaction of reducing sugars with proteins, lipids and nucleic acids. Diet has been recognized as an important exogenous source of AGEs. There is evidence for the implication of AGEs in the pathogenesis of diabetes-related complications, atherosclerosis, ageing processes or Alzheimer´s disease. Although, only little information exists about their effects in humans. The hypotheses of this study are that a high-AGE meal leads to a more important acute vascular dysfunction comparing to a low-AGE meal, and that a 1050mg/day Benfotiamine therapy for 3 days has a protective effect on the endothelial function.

Twenty-one people with type 2 diabetes shall be investigated in a randomized, single-blinded (investigator), cross-over design (please compare design description).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* age: 35-70 years

Exclusion Criteria:

* Heart failure corresponding to NYHA- class III and IV
* history of stroke
* history of myocardial infarction
* unstable angina pectoris
* peripheral artery disease stadium IIb and more
* kidney disease (Creatinine > 1,8 mg/dl and/or creatinine clearance <50 ml/min calculated according to the Cockroft formula and/or macroalbuminuria >200 mg/l)
* malignant diseases
* chronical alcohol consumption (more than 50 ml of highly concentrated alcohol or equivalents / day)
* pregnancy or lactation
* potentially child- bearing women without sufficient contraception (sufficient contraception is defined as the use of a contraceptive method that has an efficiency of over 99% (according to CHMP/EWP/225/02)). A pregnancy test will be performed before the commencement of the study.
* arterial hypotonia (blood pressure<90/50 mmHg) or arterial hypertonia with systolic blood pressure >159 mmHg and/or diastolic blood pressure >99 mmHg
* arterial hypertonia requiring more than three antihypertensive agents
* advanced diabetes complications (subjects must have been investigated with regard to these complications maximum 6 months previously by a specialized physician) such as:
* proliferative diabetic retinopathy
* diabetic neuropathy requiring morphium derivatives
* patients with an acute foot syndrome
* HbA1c >10 %
* participation to other studies within the previous 3 months

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2004-11; Study Completion 2006-01

PRIMARY OUTCOMES:
A high-AGE meal causes a more pronounced postprandial endothelial dysfunction comparing to a low-AGE meal in people with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
The influence of high-AGE vs. low-AGE meal on the laboratory parameters that mirror AGE-metabolism, oxidative stress, endothelial dysfunction and inflammation shall be investigated.
To investigate whether treatment with Benfotiamine 1050mg/day for 3 days has a protective effect on endothelial function after a high-AGE meal

CONTACTS AND LOCATIONS:
Overall Officials: Alin O Stirban, Dr, Principal Investigator — Heart and Diabetes Center NRW
Locations (1):
- Heart and Diabetes Center NRW, Bad Oeynhausen, Germany